CLINICAL TRIAL: NCT04627909
Title: Emotional Support of a Social Robot at the Pediatric Emergency Department: a Randomized Clinical Trial
Brief Title: Robot Therapy in Pediatric Emergency
Status: Completed | Type: Observational
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Clara Balsano, Ordinary professor, University of L'Aquila
Other Study IDs: prot. N. 2666 06-25-2019
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Child, Only
MeSH Terms: interventions — Health Personnel; Caregivers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group under Robot treatment: Interaction with the Humanoid Robot for 15 minutes
  Interventions: Other: Robot
- Group involved with medical personnel: Interaction with medical personnel for 15 minutes
  Interventions: Other: Medical Personnel
- Control group: Exclusive interaction with the caregiver for 15 minutes
  Interventions: Other: Caregiver

INTERVENTIONS:
Other: Robot — The patient interacts with a robot
  Groups: Group under Robot treatment
Other: Medical Personnel — The patient interacts with medical personnel
  Groups: Group involved with medical personnel
Other: Caregiver — The patient interacts with the caregiver
  Groups: Control group

SUMMARY:
The investigators are evaluating if the use of humanoid robots is an optimal distraction strategy in order to produce positive emotional states and facilitate the diagnosis and to reduce treatment time in pediatric age in emergency situations.

ELIGIBILITY:
Inclusion Criteria:

* children between the ages of 3 and 10 with white, green and yellow triage code

Exclusion Criteria:

* Red triage code
* inadequate knowledge of the Italian language,
* yellow triage code in case of: headache for recent trauma with visual impairment; headache with neck rigidity or vomiting; indifference to the environment; dyspnea and increased respiratory work; intoxication by inhalation of toxic substances; significant trauma to the head with altered state of consciousness.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children in pediatric emergency department
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol level | The surveys have been made when children arrived, after their assigned 15-minutes interaction, and twenty minutes before medical physical examination.
  The children's salivary cortisol production was measured over time to obtain a clear picture of the trend of the children's stress level before the emergency medical procedures.

SECONDARY OUTCOMES:
Psychological tests | The surveys have been made after a 15-minute interaction with the robot or mother or medical staff.
  The secondary endpoint was to explore whether and how psychological characteristics of the children, such as temperament and understanding of emotions, affected their emotional responses

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, Italy

REFERENCES:
- [Derived] Rossi S, Santini SJ, Di Genova D, Maggi G, Verrotti A, Farello G, Romualdi R, Alisi A, Tozzi AE, Balsano C. Using the Social Robot NAO for Emotional Support to Children at a Pediatric Emergency Department: Randomized Clinical Trial. J Med Internet Res. 2022 Jan 13;24(1):e29656. doi: 10.2196/29656. PMID 34854814